CLINICAL TRIAL: NCT05318456
Title: A Randomized, Triple-blind, Placebo-controlled, Parallel Clinical Trial to Investigate the Safety and Efficacy of MoodElite T-4003-1 on Improving Mood in a Healthy Adult Population With Mild to Moderate Depressive Symptoms Not Eligible for Therapeutic Intervention
Brief Title: The Safety and Efficacy of MoodElite T-4003-1 on Improving Mood in a Healthy Adult Population With Mild to Moderate Depressive Symptoms Not Eligible for Therapeutic Intervention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chenland Nutritionals Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21CNCFT01
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Mood
Keywords: Mild to moderate depression; Mild to moderate depressive symptoms not eligible for therapeutic intervention; MoodElite T-4003-1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MoodElite T-4003-1 (Experimental): Participants will be instructed to take two capsules of MoodElite T-4003-1 once daily with water, after dinner without food starting on Day 0 for 42 days. If a dose is missed participants are instructed to take the dose as soon as they remember. Participants will be advised not to exceed 4 capsules daily.
  Interventions: Dietary Supplement: MoodElite T-4003-1
- Comparator (Active Comparator): Participants will be instructed to take two capsules of comparator once daily with water, after dinner without food starting on Day 0 for 42 days. If a dose is missed participants are instructed to take the dose as soon as they remember. Participants will be advised not to exceed 4 capsules daily.
  Interventions: Dietary Supplement: Comparator
- Placebo (Placebo Comparator): Participants will be instructed to take two capsules of placebo once daily with water, after dinner without food starting on Day 0 for 42 days. If a dose is missed participants are instructed to take the dose as soon as they remember. Participants will be advised not to exceed 4 capsules daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: MoodElite T-4003-1 — Participants will be instructed to take two capsules of MoodElite T-4003-1 once daily with water, after dinner without food for 42 days.
  Arms: MoodElite T-4003-1
Dietary Supplement: Comparator — Participants will be instructed to take two capsules of comparator once daily with water, after dinner without food for 42 days.
  Arms: Comparator
Other: Placebo — Participants will be instructed to take two capsules of placebo once daily with water, after dinner without food for 42 days.
  Arms: Placebo

SUMMARY:
The objective of this study is to investigate the efficacy and safety of MoodElite T-4003-1 on improving mood in a healthy adult population with mild to moderate depressive symptoms not eligible for therapeutic intervention.

DETAILED DESCRIPTION:
The objective of this study is to investigate the safety and efficacy of 42-day supplementation of MoodElite T-4003-1 on improving mood in healthy adults. The efficacy of MoodElite T-4003-1 on mood will be assessed by the Beck Depression Inventory (BDI-II) and Profile of Mood States (POMS) Questionnaire. POMS is a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. Self-reported sleep efficiency, perceived sleep debt, and sleep difficulty will be assessed by a Sleep Quality Questionnaire and supported by sleep scoring from actigraphy readings. As vitality is related to both mood and sleep, the Vitality and Quality of Life questionnaire will be used to measure changes in energy levels and quality of life over the 42-day study period. The effects of MoodElite T-4003-1 will be compared to a placebo and comparator product, EasyMind T-4008-1. EasyMind T-4008-1 contains extracts from Paeonia lactiflora, Gardenia jasminoides, Albizia julibrissin, Paeonia suffruticosa and has been shown to reduce anxiety-like behaviour in a rodent model using chronic restraint stress through reduction of corticosterone (cortisol) (unpublished results).

For the study population, the eligibility criteria limits the presence of confounding variables that could influence study outcomes. Participants will be healthy men and women between 18 and 65 years of age. Individuals will be recruited based on having mild to moderate depressive symptoms, as assessed by the BDI-II. The BDI-II contains 21 items and evaluates both psychological and physical symptoms related to depression. Participants with diagnosed chronic or major depression or psychiatric disorders will be excluded to ensure only those with mild, non-pathological depressive symptoms are enrolled. Any participants taking prescribed or over the counter mood altering medications will be excluded, as not to interfere with the evaluation of the effects of MoodElite T-4003-1 on mood. Participants taking supplements for mood support at a stable dose for at least three months will be evaluated by the QI to determine eligibility. Shift workers or individuals who have recently travelled across one or more time zones will be excluded to limit any confounding effects on outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 18-65 years of age, inclusive
2. Individual is not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least one year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
3. Individuals with mild to mild-moderate depressive symptoms, as determined by a score of 14-24 on the BDI-II at screening, and as assessed by the Qualified Investigator (QI)
4. Education level no less than that of primary school
5. Individuals who can read and write in English and can understand the BDI-II
6. Agrees to maintain current lifestyle habits as much as possible throughout the study depending on your ability to maintain the following: diet, medications, supplements, exercise, and sleep and avoid taking new supplements during the study period
7. Provided voluntary, written, informed consent to participate in the study
8. Healthy as determined by medical history and laboratory results as assessed by QI

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients
3. History of diagnosed chronic or major depression as assessed by the QI
4. Participants undergoing behavioural therapy for depression. Participants who have completed at least 8 sessions of behavioural therapy with no improvement will be considered by the QI
5. Suicidal ideation as assessed by the BDI-II
6. History of psychiatric disorders such as organic brain disorders, bipolar affective disorder, personality disorder, as assessed by the QI
7. Diagnosed insomnia or other sleep disorders as assessed by the QI
8. Current employment that calls for shift work or have worked shift work in the last 3 weeks
9. Travel across 1 or more-time zones in the last 2 weeks and/or is anticipating more travel
10. Current use of prescribed medications, over-the-counter (OTC) medications, or supplements taken for treatment of depression or used to help sleep
11. Current use of prescribed medications that interact with Hypericum perforatum
12. Unstable metabolic disease or chronic diseases as assessed by the QI
13. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
14. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
15. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
16. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
17. Use of medical cannabinoid products
18. Current chronic use of cannabinoid products (>8 times/month) and is unwilling to stop for the duration of the study beginning 1 week prior to baseline. History of chronic and occasional use and the purpose of use to be assessed by QI on a case-by-case basis
19. Alcohol intake >2 standard drinks per day as assessed by the QI
20. Alcohol or drug abuse within the last 12 months
21. Clinically significant abnormal laboratory results at screening as assessed by the QI
22. Participation in other clinical research studies 30 days prior to enrollment will be assessed on a case-by-case basis by the QI
23. Individuals who are unable to give informed consent
24. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Change in mood between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by BDI-ll | Days 0, 42 and day 56 (follow-up)
  The change in mood between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using Beck Depression Inventory-II (BDI-II). The BDI-II contains 21 items on a 4-point scale from 0 'Symptom Absent' to 3 'Severe Symptom'. Scoring is achieved by adding the highest ratings for all 21 items with a minimum score of 0 and maximum score of 63. A higher total BDI-II score indicates greater symptom severity.
Change in total mood disturbance between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by POMS Questionnaire | Days 0, 42 and day 56 (follow-up)
  The change in total mood disturbance between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using Profile of Mood States (POMS) Questionnaire. The POMS questionnaire is used to measure mood states, with its validity well established as its methodology has been used in many clinical trials. POMS are a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. Each item contains a 5-point Likert scale characterizing the possible strengths of a specific feeling (e.g. friendly, sad, helpful) ranging from 'Not at all' to 'Extremely'.

SECONDARY OUTCOMES:
Change in tension-anxiety between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by POMS | Days 0, 42 and day 56 (follow-up)
  The change in POMS subscale of tension-anxiety between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using Profile of Mood States (POMS) Questionnaire. The POMS questionnaire is used to measure mood states, with its validity well established as its methodology has been used in many clinical trials. POMS are a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. Each item contains a 5-point Likert scale characterizing the possible strengths of a specific feeling (e.g. friendly, sad, helpful) ranging from 'Not at all' to 'Extremely'.
Change in depression between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by POMS | Days 0, 42 and day 56 (follow-up)
  The change in POMS subscale of depression between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using Profile of Mood States (POMS) Questionnaire. The POMS questionnaire is used to measure mood states, with its validity well established as its methodology has been used in many clinical trials. POMS are a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. Each item contains a 5-point Likert scale characterizing the possible strengths of a specific feeling (e.g. friendly, sad, helpful) ranging from 'Not at all' to 'Extremely'.
Change in anger-hostility between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by POMS | Days 0, 42 and day 56 (follow-up)
  The change in POMS subscale of anger-hostility between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using Profile of Mood States (POMS) Questionnaire. The POMS questionnaire is used to measure mood states, with its validity well established as its methodology has been used in many clinical trials. POMS are a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. Each item contains a 5-point Likert scale characterizing the possible strengths of a specific feeling (e.g. friendly, sad, helpful) ranging from 'Not at all' to 'Extremely'.
Change in vigor between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by POMS | Days 0, 42 and day 56 (follow-up)
  The change in POMS subscale of vigor between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using Profile of Mood States (POMS) Questionnaire. The POMS questionnaire is used to measure mood states, with its validity well established as its methodology has been used in many clinical trials. POMS are a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. Each item contains a 5-point Likert scale characterizing the possible strengths of a specific feeling (e.g. friendly, sad, helpful) ranging from 'Not at all' to 'Extremely'.
Change in fatigue between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by POMS | Days 0, 42 and day 56 (follow-up)
  The change in POMS subscale of fatigue between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using Profile of Mood States (POMS) Questionnaire. The POMS questionnaire is used to measure mood states, with its validity well established as its methodology has been used in many clinical trials. POMS are a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. Each item contains a 5-point Likert scale characterizing the possible strengths of a specific feeling (e.g. friendly, sad, helpful) ranging from 'Not at all' to 'Extremely'.
Change in confusion between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by POMS | Days 0, 42 and day 56 (follow-up)
  The change in POMS subscale of confusion between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using Profile of Mood States (POMS) Questionnaire. The POMS questionnaire is used to measure mood states, with its validity well established as its methodology has been used in many clinical trials. POMS are a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. Each item contains a 5-point Likert scale characterizing the possible strengths of a specific feeling (e.g. friendly, sad, helpful) ranging from 'Not at all' to 'Extremely'.
Change in subjective sleep efficiency between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by the Sleep Quality Questionnaire | Days 0 and 42
  The change in subjective sleep efficiency between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using the Sleep Quality Questionnaire. Participants will be asked a total of 18 questions. Four will capture information regarding a typical 7-day period consisting of 5 weekdays and 2 weekend days. The remaining 14 questions use a 5-point Likert scale ranging from 'Strongly Disagree' to 'Strongly Agree'.
Change in perceived sleep debt between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by the Sleep Quality Questionnaire | Days 0 and 42
  The change in perceived sleep debt between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using the Sleep Quality Questionnaire. Participants will be asked a total of 18 questions. Four will capture information regarding a typical 7-day period consisting of 5 weekdays and 2 weekend days. The remaining 14 questions use a 5-point Likert scale ranging from 'Strongly Disagree' to 'Strongly Agree'.
Change in perceived sleep difficulty between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by the Sleep Quality Questionnaire. | Days 0 and 42
  The change in perceived sleep difficulty between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using the Sleep Quality Questionnaire. Participants will be asked a total of 18 questions. Four will capture information regarding a typical 7-day period consisting of 5 weekdays and 2 weekend days. The remaining 14 questions use a 5-point Likert scale ranging from 'Strongly Disagree' to 'Strongly Agree'.
Change in objective sleep measures between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by actigraphy readings | Days 0 and 42
  The change in objective sleep measures between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using actigraphy readings. The actigraphy device is an objective measure of sleep during the study period. Each subject will wear the actigraphy device on their non-dominant arm for seven consecutive days prior to each study visit, allowing for charging and periods when the device is may not be worn (i.e. showering). The actigraphy device will be used to collect sleep outcome variables including but not limited to sleep start and end, average length and number of awakenings, sleep efficiency, sleep latency, time asleep, wake episodes, and fragmentation index.
Change in vitality throughout the day between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation as assessed by Vitality and Quality of Life Questionnaire | Days 0 and 42
  The change in vitality throughout the day between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be assessed using the Vitality and Quality of Life Questionnaire. The Vitality and QoL Questionnaire will be used to assess the energy levels and quality of life of the participants. The 31-item questionnaire consists of a 7-point Likert scale, with answers ranging from 1 to 7. The higher the summative score the more vitality that was subjectively perceived by the participants.
Change in blood melatonin levels between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation | Days 0 and 42
  The change in blood melatonin levels between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be measured.
Change in fecal microbiome between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation | Days 0 and 42
  The change in fecal microbiome between MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo from baseline to day 42 after supplementation will be measured.

OTHER OUTCOMES:
Incidence of pre-emergent adverse events following 42 days of supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Incidence of pre-emergent adverse events following 42 days of supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Incidence of post-emergent adverse events following 42 days of supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Incidence of post-emergent adverse events following 42 days of supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in Aspartate Aminotransferase levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo | Days 0 and 42
  Change in Aspartate Aminotransferase levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo will be determined.
Change in alanine aminotransferase levels from baseline to baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo | Days 0 and 42
  Change in alanine aminotransferase levels from baseline to baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), and placebo will be determined.
Change in urinalysis levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in urinalysis levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in alkaline phosphatase levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in alkaline phosphatase levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in total bilirubin levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in total bilirubin levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in creatinine levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in creatinine levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in potassium levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in potassium levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in sodium levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in sodium levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in chloride levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in chloride levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in glucose levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in glucose levels from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in estimated glomerular filtration rate (eGFR) from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in estimated glomerular filtration rate (eGFR) from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in white blood cell count from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in white blood cell count from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in levels of neutrophils from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in levels of neutrophils from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in levels of lymphocytes from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in levels of lymphocytes from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in levels of monocytes from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in levels of monocytes from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in levels of eosinophils from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in levels of eosinophils from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in levels of basophils from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in levels of basophils from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in levels of hemoglobin from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in levels of hemoglobin from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in levels of hematocrit from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in levels of hematocrit from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in Red Blood Cell Count from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in Red Blood Cell Count from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in platelet count from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in platelet count from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in levels of immature granulocytes from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in levels of immature granulocytes from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in levels of nucleated red blood cells from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in levels of nucleated red blood cells from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in mean corpuscular volume from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in mean corpuscular volume from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in mean corpuscular hemoglobin from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in mean corpuscular hemoglobin from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in mean corpuscular hemoglobin concentration from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in mean corpuscular hemoglobin concentration from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.
Change in red cell distribution width from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo | Days 0 and 42
  Change in red cell distribution width from baseline to 42 days following supplementation with MoodElite T-4003-1, comparator (EasyMind T-4008-1), or placebo will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada